CLINICAL TRIAL: NCT01515813
Title: A Randomized Controlled Trial to Compare the Effects of Highly Active Antiretroviral Therapy (HAART) Versus Statin Therapy on Endothelial Function and Markers of Inflammation/Coagulation In HIV-Infected Individuals With High CD4 Cell Counts
Brief Title: Effect of HAART Vs. Statin Treatment on Endothelial Function and Inflammation/Coagulation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: On 05/08/12, team working on revising protocol and re-open study under version 2.0
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5292; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-11-08; First posted 2012-01-24 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Pravastatin; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Pravastatin sodium alone for 24 weeks (Experimental): One 40 mg tablet of Pravastatin sodium taken orally once daily for 24 weeks starting at week 0 and ending at week 24.
  Interventions: Drug: Pravastatin sodium
- Arm B: EFV/FTC/TDF plus Pravastatin sodium at week 13 (Experimental): EFV/FTC/TDF once daily for 24 weeks starting at week 0 and ending at week 24 plus pravastatin sodium (80 mg)once daily for 12 weeks starting at week 13 ending at week 24.
  Interventions: Drug: Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate; Drug: Pravastatin sodium
- Arm C: Pravastatin sodium + EFV/FTC/TDF for 24 weeks (Experimental): Participants will be administered Pravastatin sodium once daily for 24 weeks starting at week 0 and ending at week 24 plus EFV/FTC/TDF once daily for 24 weeks starting week 0 and ending at week 24.
  Interventions: Drug: Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate; Drug: Pravastatin sodium

INTERVENTIONS:
Drug: Pravastatin sodium — One 40 mg tablet of Pravastatin sodium taken orally once daily.
  Arms: Arm A: Pravastatin sodium alone for 24 weeks
Drug: Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate — Participant will be administered one tablet of Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF)600 mg/200 mg/300 mg taken orally once daily
  Other Names: EFV/FTC/TDF
  Arms: Arm B: EFV/FTC/TDF plus Pravastatin sodium at week 13; Arm C: Pravastatin sodium + EFV/FTC/TDF for 24 weeks
Drug: Pravastatin sodium — Two 40mg tablets (80 mg total) of Pravastatin sodium taken orally once daily.
  Arms: Arm B: EFV/FTC/TDF plus Pravastatin sodium at week 13; Arm C: Pravastatin sodium + EFV/FTC/TDF for 24 weeks

SUMMARY:
Since people started taking HIV medications, illnesses related to AIDS have decreased, but other serious illnesses like heart disease (heart attacks) and certain kinds of cancer have increased. Studies show that HIV causes changes in the lining of the arteries and also causes inflammation (irritation) inside the body that may play a role in diseases like heart attacks and strokes. The levels of inflammation and artery lining health can also affect how well your brain works. These changes cannot be felt, but can be measured. Artery lining health can be looked at with a test that uses a blood pressure cuff on your arm to see how the artery responds when air is let in and out of the cuff. An ultrasound (machine that uses sound waves) is used to look at the artery during the test. This test is called Flow Mediated Dilation or FMD for short. Inflammation can be checked with blood tests (blood tests that measure this irritation inside the body that you cannot feel). HIV medications can improve the artery lining health and can partially lower levels of inflammation in the blood; however, these levels of inflammation may not be able to return back to normal.

Pravastatin sodium is a medication that is approved by the Food and Drug Administration (FDA) for treating high cholesterol. Pravastatin sodium has also been able to improve the health of the lining of the arteries and lower the level of inflammation in people with other diseases, but has not been studied or approved for this purpose in people who have HIV. This research study will look at the effects of two types of medications used separately or together on the health of the lining of arteries and levels of inflammation in the blood: Atripla (a HIV medication) and pravastatin sodium. This study will also look at the effects of Atripla and pravastatin sodium on cholesterol levels, tests that measure how well you can think and calculate (tests of neurocognitive function), and at the effects of Atripla on the levels of pravastatin sodium in the blood.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Willingness to defer initiation of ART for up to 24 weeks or statin therapy for up to 12 weeks after study entry.
* CD4+ cell count >500/mm3 within 60 days prior to study entry obtained at any laboratory that has a CLIA certification or its equivalent.
* No prior ART of more than 10 cumulative days with the following exceptions:

  * Use of ART drugs as part of post-exposure prophylaxis (PEP) provided the participant did not acquire HIV-1 infection from the event that required PEP.
  * ART use during pregnancy that resulted in virologic suppression based on the assay available at the time and was not complicated while on therapy either by detectable HIV-1 RNA following suppression or the development of resistance. Women who received ZDV monotherapy prior to the availability of viral load testing will still be considered eligible as long as ZDV was not taken for more than 12 weeks. ART must have been stopped within 4 weeks of delivery and cannot have been received within 6 months of the A5292 screening visit.
  * Receipt of ARV drugs while HIV-uninfected, with documentation of negative HIV-1 serology at least 90 days after completion of ARV drugs.
* No lipid-lowering medication (prescription or non-prescription) within 60 days prior to study entry. This includes all statin drugs, omega-3-fatty acids/fish oil (if dose > 1 g/day), red yeast rice (any dose), and niacin products (e.g., niacin, nicotinic acid, vitamin B3; if dose of >100 mg/day), in addition to those listed on the A5292 PSWP.
* No ART within the past 30 days.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* In the opinion of the investigator, no medical, mental health or other condition that precludes participation.
* Certain laboratory values obtained within 60 days prior to entry, as indicated in section 4.1.10 of the protocol.
* Framingham Risk Score (FRS) greater than/equal to 10% OR FRS greater than/equal to 6% if hsCRP > 3.0 mg/L OR participant has controlled type ll diabetes mellitus.
* No evidence of any exclusionary resistance mutations based on results from any genotype assay from any laboratory that has a CLIA certification or its equivalent. The result must either be available from previous testing or must be obtained prior to entry and have been reviewed by the site investigator. If a genotype is submitted, but for technical reasons cannot be completed, the participant will still be allowed to enroll, if otherwise eligible. (The protocol will not provide the resistance assay). An exclusionary resistance mutation is defined in section 4.1.12 of the protocol.
* Completion of the pre-entry FMD assessment.
* For women of reproductive potential, negative serum or urine pregnancy test with a sensitivity of ≤ 25 mIU/mL at screening and within 72 hours prior to study entry.
* Female study volunteers of reproductive potential include women who have not been post-menopausal for at least 24 consecutive months, (i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy).
* Contraception requirements-

  * All subjects must agree not to participate in the conception process and if participating in sexual activity that could lead to pregnancy, must agree to use at least two reliable methods of contraception for 2 weeks before study treatment, while receiving study treatment, and for 6 weeks after receiving study treatment. As hormone-based contraceptives can affect coagulopathy biomarkers, subjects who plan on using such a contraceptive during the study must be taking the same product for at least 30 days prior to screening and be encouraged to continue throughout the duration of the study, if medically feasible.
  * Subjects receiving an EFV-based regimen must use a barrier method as one of the two forms of contraception. Acceptable types of contraception include male or female condoms (with or without a spermicidal agent), diaphragm or cervical cap with spermicide, intrauterine device (IUD), and hormone-based contraceptive
* Female subjects who are not of reproductive potential or whose male partner(s) has azoospermia are eligible to start study drugs without requiring the use of contraceptives. Confirmation of the lack of reproductive potential is REQUIRED and written documentation or oral communication from a clinician or clinician's staff must be documented in source documents of either a physician report/letter, operative report or other source documentation in the patient record, discharge summary, laboratory report of azoospermia, or FSH measurement elevated into the menopausal range as established by the reporting laboratory.
* Ability and willingness to complete the neuropsychological tests.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
* Known and documented cardiovascular disease (history of MI, coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, peripheral arterial disease with ABI <0.9 or claudication).
* Uncontrolled type II diabetes mellitus.
* History of hepatic cirrhosis.
* Known chronic inflammatory conditions such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, sarcoidosis, inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis), chronic pancreatitis, or autoimmune hepatitis, myositis, or myopathy.
* Known active or recent (not fully resolved within 30 days prior to study entry) systemic bacterial, fungal, parasitic, or viral infections.
* Serious illness or trauma requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
* Febrile (temperature >100.4 F [38 C]) or acute illness on the day the initial study FMD is performed.
* Current severe congestive heart failure (New York Heart Association [NYHA] Class III or IV). See A5292 MOPS for stages of heart failure.
* Uncontrolled hypertension within 60 days prior to study entry (systolic > 160 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings on two or more occasions. NOTE: If the initial blood pressure reading is >160 mm Hg (systolic) or > 100 mm Hg (diastolic), then the participant must come back to the clinic for additional readings prior to study entry.
* Documented untreated hypothyroidism per participant's medical records. Subjects with treated hypothyroidism are allowed. NOTE: A thyroid stimulating hormone evaluation is not required by this study.
* Current use of thyroid hormone supplements (e.g., levothyroxine, liothyronine, thyroid extract) other than for treatment of hypothyroidism.
* Active cancer requiring systemic chemotherapy or radiation.
* Active brain infection, brain neoplasm, or space-occupying brain lesion requiring acute, or chronic therapy. Subjects with active fungal meningitis, toxoplasmosis, or CNS lymphoma are excluded from participation.
* Not fasting (see Section 6.3.1 of the protocol) or refraining from smoking or exercising for the 8 hours prior to evaluations on the day of pre-entry FMD assessment. Refer to A5292 MOPS for complete instructions.
* At the time of study entry planning to start or stop smoking during the first 12 weeks of the trial.
* At the time of study entry planning to initiate chronic therapy with anti-inflammatory agents (such as aspirin) or immunomodulators during the first 12 weeks of the trial.
* At the time of study entry planning to significantly change diet or exercise habits during the study period.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any active psychiatric illness including schizophrenia, severe depression, or severe bipolar affective disorder that, in the opinion of the investigator, could confound the analysis of the neurological examination or neuropsychological test results.
* Hormonal anabolic therapies within 90 days prior to study entry including, but not limited to growth hormone (Serostim), nandrolone (Deca-Durabolin), oxandrolone (Oxandrin), oxymetholone (Anadrol-50), stanozolol (Winstrol), methyltestosterone (Oreton Methyl), fluoxymesterone (Halotestin), megestrol acetate (Megace) and tesamorelin.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational immunomodulator therapy within 60 days prior to study entry. NOTE: Routine standard of care vaccinations including hepatitis A and/or B, influenza, pneumococcal, and tetanus are permitted if administered at least 7 days before entry evaluations.
* Current use of vitamin E supplements greater than 200 IU/day.
* Current use of vitamin C supplements greater than 250 mg/day.
* Any systemic glucocorticoid above replacement levels, defined as the equivalent of > 7.5 mg of prednisone daily, within 60 days of entry. NOTE: Topical, nasal and inhaled glucocorticoid agents are permitted, provided the participant has been on stable dosage(s) for at least 30 days prior to entry and has no plans to alter dosage(s) and/or frequency during the first 12 weeks of the trial.
* Currently taking or anticipation of starting medication during the study for hepatitis C including interferon and ribavirin.
* Use of investigational therapies within 90 days prior to study entry unless approved by A5292 core team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in brachial artery FMD | From week 0 to week 12

SECONDARY OUTCOMES:
Change in IL-6 | From week 0 to week 12
Change in hs-CRP | From week 0 to week 12
Change in D-dimer | From week 0 to week 12
Change in non-HDL cholesterol | From week 0 to week 12
Change in fasting triglycerides | From week 0 to week 12
Change in demographically corrected standard scores (T-scores) for each neuropsychological performance domain and the overall global deficit score (GDS) | From week 0 to week 12
Change in brachial artery FMD | From week 0 to week 24
Change in IL-6 | From week 0 to week 24
Change in hs-CRP | From week 0 to week 24
Change in D-dimer | From week 0 to week 24
Change in non-HDL cholesterol | From week 0 to week 24
Change in fasting triglycerides | From week 0 to week 24
Change in demographically corrected standard scores (T-scores) for each neuropsychological performance domain and the overall global deficit score (GDS) | From week 0 to week 24

CONTACTS AND LOCATIONS:
Overall Officials: David A. Wohl, M.D., Study Chair — University of North Carolina AIDS CRS
Locations (9):
- United States (9):
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - Washington University CRS (2101), St Louis, Missouri
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke University Medical Center Adult CRS (1601), Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS (3203), Greensboro, North Carolina
  - The Ohio State University AIDS CRS (2301), Colombus, Ohio
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas